CLINICAL TRIAL: NCT03095261
Title: A Web-based Exercise Intervention With Financial Incentives for Cardiac Rehabilitation Graduates: A One Year Crossover Study Design
Brief Title: Incentives in Cardiac Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Paul Oh, Medical Director of the Cardiovascular Prevention and Rehabilitation Program, University Health Network, Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 15-9066
Record Dates: First submitted 2016-10-13; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular Disease; Cardiac Rehabilitation; Financial Incentives; Outpatient (Phase II) Cardiac Rehabilitation Exercise Adherence
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-monitoring (financial incentives then virtual rewards) (Experimental): Participants will be asked to track their exercise daily, using an online tool called ExTracker.ca, for 52 weeks. Date, type of exercise, time spent exercising, and distance covered will be self-reported, as will steps per day and 10-minute bouts of MVPA per day (measured by an accelerometer). In the first six months, participants will earn financial incentive (ex. grocery vouchers) each day exercise is tracked. In the second six months, participants will earn virtual rewards (i.e. heart badges) each day exercise is tracked.
  Interventions: Behavioral: Web-based exercise diary; Device: Accelerometer; Behavioral: Financial Incentive
- Self-monitoring (virtual rewards then financial incentives) (Active Comparator): Participants will be asked to track their exercise daily, using an online tool called ExTrack.ca, for 52 weeks. Date, type of exercise, time spent exercising, and distance covered will be self-reported, as will steps per day and 10-minute bouts of MVPA per day (measured by an accelerometer). In the first six months, participants will earn virtual rewards (i.e. heart badges) each day exercise is tracked. In the second six months, participants will earn financial incentive (ex. grocery vouchers) each day exercise is tracked.
  Interventions: Behavioral: Web-based exercise diary; Device: Accelerometer; Behavioral: Virtual Reward

INTERVENTIONS:
Behavioral: Web-based exercise diary — All participants will have access to a web-based exercise tracking tool called ExTracker. Individuals will be asked to submit their exercise diaries daily for 52 weeks, using the ExTracker program. Upon entering exercise information, participants will receive individual (e.g., You've completed 50% of your exercise sessions this week!) and group-level (e.g., You and the other people in this study are walking across Canada! Next stop - Toronto!) feedback. Should participants cease to use the platform for one week, they will receive an email reminder to re-engage with the platform. Three such emails will be sent to lapsing participants.
Device: Accelerometer — All participants will be asked to wear the StepsCount Piezo accelerometer, and track the steps per day and bout minutes of MVPA per day measured by the device. Additionally, participants will be mailed an accelerometer (and asked to return their used ones) at study weeks 26 and 52 in order for the researcher to confirm the data inputted into the ExTracker from the device.
Behavioral: Virtual Reward — Participants will earn 'virtual rewards' (i.e. a heart badge) each day they track their exercise, for the first six months of the study. In the second six months, participants will "crossover" to the other therapy, the 'financial incentive' therapy, for six months.
  Arms: Self-monitoring (virtual rewards then financial incentives)
Behavioral: Financial Incentive — Participants will earn financial incentives each day they track their exercise, for the first six months of the study. In the second six months, participants will "crossover" to the other therapy, the 'virtual rewards' therapy, for six months.
  Arms: Self-monitoring (financial incentives then virtual rewards)

SUMMARY:
The objective of this study is to examine whether a financial incentive program increases minutes of moderate-to-vigorous physical activity (MVPA) per week among cardiac rehabilitation (CR) graduates.

DETAILED DESCRIPTION:
A 52-week, randomized, crossover study design will be employed to examine the impact of financial incentives on MVPA among cardiac rehabilitation (CR) program graduates. Two experimental therapies, (1) online self-monitoring plus 'virtual rewards' (i.e. badges) (ExTrack.ca) and (2) online self-monitoring plus 'financial incentives' (ExTracker.ca), will be administered for six months, one after the other.

Study participants will be randomly assigned (1:1) to receive these therapies in one of two orders: Group A will receive ExTrack.ca (virtual rewards) for six months, followed by ExTracker.ca (financial incentives) for the next six months; Group B will receive the financial incentive condition first, and the virtual rewards condition second. While exposed to the incentive condition, participants will be eligible to earn financial reward per day exercise is tracked.

This study design allows for the assessment of 'real world' uptake of an incentive program among CR patients, since both Groups A and B will be able to earn incentives. This design will also help determine if incentives sustain MVPA in the first six months post-CR compared with the virtual rewards condition. Finally, the crossover design will allow the exploration of incentive 'timing' - that is, figuring out if incentives more effectively sustain MVPA post-CR if they are offered immediately, versus six months after graduation when patient motivation tends to wane.

In addition to tracking exercise sessions using the online self-monitoring tool, participants will be asked to record steps per day, and 10-minute MVPA bouts per day, using a StepsCount accelerometer. To check the accuracy of participant entries, participants will be asked to mail-in their accelerometers at the study mid- and end-points (26 and 52 weeks, respectively). Participants will also be asked to complete the Behavioural Regulation to Exercise Questionnaire (BREQ-3) at baseline (T1), study mid-point/crossover (T2), and study end-point (T3) as well as cardiopulmonary fitness assessments at T1 and T3.

ELIGIBILITY:
Inclusion Criteria:

* CR program graduate (actively participating in program in month six, the final month, of the CR program).

Exclusion Criteria:

* No internet access
* Non-English speaking
* Diagnosed cognitive disorder
* Participating in another post-CR intervention study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in minutes of objectively measured moderate to vigorous intensity physical activity (MVPA) at 6 months | Baseline and 6 months
  The primary outcome of this trial will be minutes of objectively assessed MVPA per week measured by StepsCount Piezo accelerometers from baseline to 6 months.

SECONDARY OUTCOMES:
Change from 6 months (intervention end) in minutes of objectively measured MVPA at 12 months | 6 months and12 months
  MVPA minutes per week from 6 months to 12 months will be a secondary outcome.
Change from baseline in Aerobic fitness at 12 months | Baseline and12 months
  Aerobic fitness will be a secondary outcome as well, measured by symptom limited exercise stress test at baseline and 12 months, given its strong and graded (inverse) associations with cardiovascular disease-related outcomes.

OTHER OUTCOMES:
Change from baseline in Motivation at 6 months and 12 months | Baseline, 6 months and12 months
  Participants will also be asked to complete a 23-item questionnaire designed to measure self-determined motivation to exercise (the BREQ-3) (Wilson et al. 2006) at Baseline, 6 months, and 12 months.
Enrolment | 12 months
  Study recruitment rate will be calculated by dividing the number of consenting CR patients by the number of eligible CR graduates who were recruited to participate in the study.
Engagement | 12 months
  Level of engagement will be defined as proportion of days ExTracker data submitted.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Oh, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Rehabilitation Insitute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No